CLINICAL TRIAL: NCT03383549
Title: Home-rehabilitation Protocol in Elderly Subjects With Mild Cognitive Impairment (MCI) Based on Information and Communications Technology (ICT) and Serious Games for Cognitive and Physical Training. Games for Older Adults Active Life (GOAL)
Brief Title: Cognitive and Physical Home-rehabilitation by Information and Communications Technology. Games for Older Adults Active Life (GOAL)
Acronym: GOAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Consorzio di Bioingeneria e Informatica Medica (Unknown); University of Florence (Other); Gutenberg Srl (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DongnocchiGOAL
Record Dates: First submitted 2017-12-15; First posted 2017-12-26 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Cognitive Dysfunction; Mild Cognitive Impairment; Vascular Cognitive Impairment
Keywords: Telerehabilitation [E02.831.891]; Cognitive Aging [G07.345.124.260]; Exercise Therapy [E02.760.169.063.500.387]
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-rehabilitation (Experimental): Tele-rehabilitation arm undergo a home-based rehabilitation combined protocol, made up of cognitive and physical exercises
  Interventions: Other: Tele-rehabilitation
- Control group (No Intervention): Control group receives only verbal instructions to train cognitive and physical conditions. Instructions will aim to promote daily and leisure activities.

INTERVENTIONS:
Other: Tele-rehabilitation — Each subject undergoes a combined rehabilitation protocol, which will be administered on a daily basis, designed to alternate physical exercises and cognitive training. Each daily session lasts between 30 and 45 minutes. The complete protocol lasts 8 weeks.
  Arms: Tele-rehabilitation

SUMMARY:
Aging is often associated with pathological pathway such as in Mild Cognitive Impairment (MCI), and that pathway may be associated to a high risk of dementia.

Tools for early identification of functional and cognitive decline and effectiveness of treatments in counteracting the loss of functionality to preserve MCI subjects autonomy, have been widely debated in recent years.

In literature, the importance of combined cognitive and physical training is also recognized (Karssemeijer E, 2017).

Moving from the above mentioned findings and considerations, the aim of GOAL project is to test a newly developed tele-rehabilitation platform to monitor and preserve functional and cognitive abilities in individuals affected by Mild Cognitive Impairment (MCI).

Participants will be enrolled and randomly assigned to the tele-rehabilitation (GOAL group) or usual care program (control group). A dedicated application will be developed for the GOAL group. Thanks to the application, the participant will access different contents, such as serious games to train cognitive abilities (Anguera et al,2013) and physical training video lessons to endorse daily activity. Each participant of GOAL group will be provided with a tablet, with the application installed on it, and an internet connection (if needed).

DETAILED DESCRIPTION:
30 patients will be allocated in the treatment arm (Telerehabilitation program, GOAL group) by randomization. Randomization will be applied with a ratio of 1:1.

The Telerehabilitation program is conceived as a combined protocol to train both cognitive and physical domains. Participants will be requested to perform the cognitive training three times weekly and physical training two times weekly, on alternate days. The subject will access the Telerehabilitation contents by using a web application configured on a touchscreen notebook, that will be provided to each participant by the research institute.

Physical exercises are going to be chosen according to adaptive physical activity model, and each session will be made up of eleven exercises, divided in three categories: warm-up, strengthening and stretching/relaxation. The participants will perform the exercises according to instructions received in a sequence of videos. Every session will last 30 minutes.

Cognitive training will be based on BrainHQ exercises (BrainHQ, Posit Science,USA) which are characterized by adaptive control of the difficulty levels. The chosen exercises aim to train different cognitive domains including: attention, executive function, memory, processing speed, reasoning, and visuospatial memory. Each session will last 20 minutes, and will include four different types of exercise.

While enrolled in the 8 weeks program, participants will also be requested to wear an actigraph. The actigraph will be placed on the non-dominant arm and will be used to monitor daily activity and sleep quality.

At the end of the tele-rehabilitation program, participants will undergo a final assessment.

ELIGIBILITY:
Inclusion criteria:

* Age between 65 and 80 years old
* Agreement to participate, with signature of the informed-consent form
* Availability of a caregiver/study partner, who agrees to support the participant through the GOAL program. Participant and caregiver are not required to live together
* Mini Mental State Examination (MMSE) score >24 The participant should present a mild cognitive impairment (MCI) in absence of secondary causes of dementia (hypothyroidism untreated or treated with a therapy that has been revised in the previous 6 months, vitamin B12 or folate deficiency), assessed through a blood test.

In case of MCI due to Alzheimer Disease (AD), additional inclusion criteria are:

* Hachinski Ischemic Score ≤4
* Absence of secondary causes of dementia confirmed by a neuroimaging examination (TC scan or encephalic MRI), Fazekas score <2
* Biomarker of neuronal damage (PET with 18f-fluorodeoxyglucose, MRI with hippocampal volumetric assessment or levels of t-tau and p-tau in the cerebrospinal fluid) or biomarkers of Aβ deposition (Amyloid-PET or levels of A> 42 in the cerebrospinal fluid) consistent with MCI due to AD

In case of MCI due to Vascular Cognitive Impairment, additional inclusion criteria are:

* Hachinski Ischemic score > 4
* Fazekas score >=2
* Presence of at least one of the following conditions, as assessed by TC scan or encephalic MRI

  * Multiple lesions in the white matter consistent with cerebral small vessel disease
  * Lacunar status
  * Multi-infarct encephalopathy with ischemic multiple lesions in the cortical region, in the basal ganglia and white matter

Exclusion Criteria:

* Unreliable communication (eg, foreign language or aphasia)
* Severe visual or auditory deficit, not reversible, to the extent that it compromises the interaction with the operator and the usage of ICT instrumentation.
* Presence of neurological and/or psychiatric disorders (Hamilton scale >12) that might interfere with cognitive status
* Left-handed individuals
* Level of education <3 years
* History of substance abuse (nicotine excluded)
* Having relapsing systemic disease and presence of major head trauma

  * Frank dementia
  * MMSE <24

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Comparison between the cognitive ability measured at the end of the treatment (time point 2 months) and at the screening time point | At the screening time point and after 2 months of treatment
  Changes in cognitive ability will be assessed by Montreal Cognitive Assessment (MoCA) Test (Conti et al., 2014)

SECONDARY OUTCOMES:
Maintenance or improvement of the physical activity | At the screening time point and after 2 months of treatment
  Physical activity performed during the trial will be evaluated through the output of the actigraph device and physical performance using the Short Physical Performance Battery
Copy and Recall of Rey's Figure | At the screening time point and after 2 months of treatment
  Copy and Recall of Rey's Figure ( Caffarra et al., 2002)
Verbal fluency task | At the screening time point and after 2 months of treatment
  Verbal fluency task (semantic - Novelli et al, 1986 - and phonemic - Carlesimo et al, 1996)
Stroop Test | At the screening time point and after 2 months of treatment
  Stroop Test (short version; Caffarra et al., 2002)
Serious Game test | At the screening time point and after 2 months of treatment
  Serious Game test (Zucchella et al, 2014)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Macchi, MD, Principal Investigator — University of Florence
Locations (1):
- Rehabilitation Centre IRCCS Don Carlo Gnocchi Foundation, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Karssemeijer EGA, Aaronson JA, Bossers WJ, Smits T, Olde Rikkert MGM, Kessels RPC. Positive effects of combined cognitive and physical exercise training on cognitive function in older adults with mild cognitive impairment or dementia: A meta-analysis. Ageing Res Rev. 2017 Nov;40:75-83. doi: 10.1016/j.arr.2017.09.003. Epub 2017 Sep 12. PMID 28912076
- [Background] Anguera JA, Boccanfuso J, Rintoul JL, Al-Hashimi O, Faraji F, Janowich J, Kong E, Larraburo Y, Rolle C, Johnston E, Gazzaley A. Video game training enhances cognitive control in older adults. Nature. 2013 Sep 5;501(7465):97-101. doi: 10.1038/nature12486. PMID 24005416
- [Background] Caffarra P, Vezzadini G, Dieci F, Zonato F, Venneri A. Rey-Osterrieth complex figure: normative values in an Italian population sample. Neurol Sci. 2002 Mar;22(6):443-7. doi: 10.1007/s100720200003. PMID 11976975
- [Background] C. Novelli, C. Papagno, E. Capitani, M. Laiacona, G. Vallar, S.F. Cappa Tre test clinici di ricerca e produzione lessicale: taratura su soggetti normalis Arch Psicol Neurol Psichiatr, 47 (1986), pp. 477-506
- [Background] Carlesimo GA, Caltagirone C, Gainotti G. The Mental Deterioration Battery: normative data, diagnostic reliability and qualitative analyses of cognitive impairment. The Group for the Standardization of the Mental Deterioration Battery. Eur Neurol. 1996;36(6):378-84. doi: 10.1159/000117297. PMID 8954307
- [Background] Zucchella C, Sinforiani E, Tassorelli C, Cavallini E, Tost-Pardell D, Grau S, Pazzi S, Puricelli S, Bernini S, Bottiroli S, Vecchi T, Sandrini G, Nappi G. Serious games for screening pre-dementia conditions: from virtuality to reality? A pilot project. Funct Neurol. 2014 Jul-Sep;29(3):153-8. PMID 25473734
- [Background] Conti S, Bonazzi S, Laiacona M, Masina M, Coralli MV. Montreal Cognitive Assessment (MoCA)-Italian version: regression based norms and equivalent scores. Neurol Sci. 2015 Feb;36(2):209-14. doi: 10.1007/s10072-014-1921-3. Epub 2014 Aug 20. PMID 25139107
- [Derived] Mosca IE, Salvadori E, Gerli F, Fabbri L, Pancani S, Lucidi G, Lombardi G, Bocchi L, Pazzi S, Baglio F, Vannetti F, Sorbi S, Macchi C. Analysis of Feasibility, Adherence, and Appreciation of a Newly Developed Tele-Rehabilitation Program for People With MCI and VCI. Front Neurol. 2020 Nov 27;11:583368. doi: 10.3389/fneur.2020.583368. eCollection 2020. PMID 33329326
- [Derived] Fabbri L, Mosca IE, Gerli F, Martini L, Pancani S, Lucidi G, Savazzi F, Baglio F, Vannetti F, Macchi C; GOAL Working Group. The Games for Older Adults Active Life (GOAL) Project for People With Mild Cognitive Impairment and Vascular Cognitive Impairment: A Study Protocol for a Randomized Controlled Trial. Front Neurol. 2019 Jan 11;9:1040. doi: 10.3389/fneur.2018.01040. eCollection 2018. PMID 30687208